CLINICAL TRIAL: NCT00495547
Title: A Multicenter, Non-Randomized, Open-Label Study to Evaluate Efficacy and Safety of Azacitidine and Beta Erythropoietin Treatment in Patients With Myelodysplastic Syndrome Red Cell Transfusion Dependent With Low or Intermediate -1 Risk.
Brief Title: SIMIDIS: Azacitidine and Beta Erythropoietin Treatment in Patients With Myelodysplastic Syndrome
Acronym: SIMIDIS
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: PETHEMA Foundation (Other)
Collaborators: Roche Pharma AG (Industry); Celgene Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2007-000972-18; SIMIDIS
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2014-04-07 (Estimated); Status verified 2014-04

CONDITIONS: Myelodysplastic Syndrome
Keywords: Myelodysplastic Syndrome; Red Cell transfusion dependent
MeSH Terms: conditions — Myelodysplastic Syndromes | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Azacitidine — Azacitidine
Drug: Beta Erythropoietin — Beta Erythropoietin

SUMMARY:
The primary objective is to evaluate the efficacy of the treatment in response rate terms. Otherwise this study wants to evaluate the safety of the treatment.

DETAILED DESCRIPTION:
A total of up to 30 patients diagnosed of myelodysplastic syndrome red cell transfusion dependent with low or intermediate -1 risk will be included.

The patients will be evaluated at scheduled visits in up to three study periods: Pre-treatment, Treatment and Follow up.

The Pre-treatment includes Screening and baseline visits. After providing informed consent, patients will be evaluated for study eligibility.

During Treatment Period patients will be evaluated once a month although biochemistry and haematology parameters will be evaluated every 2 weeks.

If an erythroid response after 24 weeks is determined, a extension treatment will be carry out without disease progression.

ELIGIBILITY:
Inclusion Criteria:

1. Must voluntary sign the informed consent.
2. Age ≥ 18 years.
3. Must be able to comply with the protocol requirements
4. Patient recently diagnosed with Myelodysplastic syndrome red cell transfusion dependent with low or intermediate -1 risk according IPSS criteria.
5. Red cell transfusion dependent anemia.
6. El patient has to be able to complain with the protocol visits.
7. Women and man must accept to use high efficacy anticonceptive methods

Exclusion Criteria:

1. Pregnancy or breast-feed women.
2. Patients previously received treatment with azacytidine .
3. Patients previously received treatment with erythropoietin agents.
4. Proliferative Chronic myelomonocytic Leukaemia (leukocytes ≥ 12000/mL).
5. Patient with a previous clinical history of another cancer (except for basocellular carcinoma or spinocellular carcinoma in situ of cervix or breast) except if the patient is free of symptoms during ≥ 3 years.
6. Cytotoxic chemotherapy or experimental agents usage for myelodysplastic syndrome treatment during 28 days.
7. Previous haematopoietic transplant.
8. Mielosupresion and antitumoral treatment during the previous 28 days.
9. The following laboratory data:

   Absolute neutrophil count < 1000 cel/ml (0.5x 109L) Platelet count < 50000/μL (25 x 109/L) Creatinine > 2.0 mg/dL (177 mmol/L) Aspartate transaminase (AST) or Alanine transaminase (ALT ) > 5 x the upper limit of normal. Total bilirubin: > 2 mg/dL
10. Patients with B12 vitamin, folic acid and ferrum deficiency.
11. Patient with positive VIH-1.
12. Any other organic or mental illness that could make impossible to sign the Inform consent or involve risk to the patient.
13. Patient has hypersensitivity previous to beta ,azacytidine, erythropoietin and/or mannitol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2009-02; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
Evaluate the efficacy of the treatment in response rate terms | 6 months

SECONDARY OUTCOMES:
Evaluate the safety of the treatment | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Sanz Guillermo, Dr, Study Director — Hospital La Fe; Del Cañizo Consuelo, DR, Study Director — Hospital Clinico de Salamanca
Locations (10):
- Spain (10):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Clínic Universitari, Barcelona
  - Hospital del Mar, Barcelona
  - Hospital Reina Sofía, Córdoba
  - Hospital Virgen Blanca, León
  - Hospital la Paz, Madrid
  - Hospital Central de Asturias, Oviedo
  - Hospital Son Llatzer, Palma de Mallorca
  - Hospital Clinico Universitario, Salamanca
  - Hospital La Fe de Valencia, Valencia

REFERENCES:
- [Background] Bennett JM, Catovsky D, Daniel MT, Flandrin G, Galton DA, Gralnick HR, Sultan C. Proposals for the classification of the myelodysplastic syndromes. Br J Haematol. 1982 Jun;51(2):189-99. PMID 6952920
- [Background] 2. Brunning RD, Head D, Bennett JM, Vardiman JW, Flandrin G, Harris NL et al. Myelodysplastic syndromes: introduction. En: Jaffe ES, Harris NL, Stein H, Vardiman JW, eds. Tumours of haematopoietic and lymphoid tissues. Lyon, IARC Press, 2001; 63-67.
- [Background] San Miguel JF, Sanz GF, Vallespi T, del Canizo MC, Sanz MA. Myelodysplastic syndromes. Crit Rev Oncol Hematol. 1996 May;23(1):57-93. doi: 10.1016/1040-8428(96)00197-7. No abstract available. PMID 8817082
- [Background] Sanz GF, Sanz MA, Vallespi T, Canizo MC, Torrabadella M, Garcia S, Irriguible D, San Miguel JF. Two regression models and a scoring system for predicting survival and planning treatment in myelodysplastic syndromes: a multivariate analysis of prognostic factors in 370 patients. Blood. 1989 Jul;74(1):395-408. PMID 2752119
- [Background] Aul C, Giagounidis A, Germing U. Epidemiological features of myelodysplastic syndromes: results from regional cancer surveys and hospital-based statistics. Int J Hematol. 2001 Jun;73(4):405-410. doi: 10.1007/BF02994001. PMID 11503953
- [Background] Sanz GF, Sanz MA, Greenberg PL. Prognostic factors and scoring systems in myelodysplastic syndromes. Haematologica. 1998 Apr;83(4):358-68. PMID 9592987
- [Background] Greenberg P, Cox C, LeBeau MM, Fenaux P, Morel P, Sanz G, Sanz M, Vallespi T, Hamblin T, Oscier D, Ohyashiki K, Toyama K, Aul C, Mufti G, Bennett J. International scoring system for evaluating prognosis in myelodysplastic syndromes. Blood. 1997 Mar 15;89(6):2079-88. PMID 9058730
- [Background] Alessandrino EP, Amadori S, Barosi G, Cazzola M, Grossi A, Liberato LN, Locatelli F, Marchetti M, Morra E, Rebulla P, Visani G, Tura S; Italian Society of Hematology. Evidence- and consensus-based practice guidelines for the therapy of primary myelodysplastic syndromes. A statement from the Italian Society of Hematology. Haematologica. 2002 Dec;87(12):1286-306. PMID 12495903
- [Background] Bowen D, Culligan D, Jowitt S, Kelsey S, Mufti G, Oscier D, Parker J; UK MDS Guidelines Group. Guidelines for the diagnosis and therapy of adult myelodysplastic syndromes. Br J Haematol. 2003 Jan;120(2):187-200. doi: 10.1046/j.1365-2141.2003.03907.x. No abstract available. PMID 12542475
- [Background] NCCN practice guidelines for the myelodysplastic syndromes. National Comprehensive Cancer Network. Oncology (Williston Park). 1998 Nov;12(11A):53-80. No abstract available. PMID 10028503
- [Background] Malcovati L, Porta MG, Pascutto C, Invernizzi R, Boni M, Travaglino E, Passamonti F, Arcaini L, Maffioli M, Bernasconi P, Lazzarino M, Cazzola M. Prognostic factors and life expectancy in myelodysplastic syndromes classified according to WHO criteria: a basis for clinical decision making. J Clin Oncol. 2005 Oct 20;23(30):7594-603. doi: 10.1200/JCO.2005.01.7038. Epub 2005 Sep 26. PMID 16186598
- [Background] Cheson BD, Bennett JM, Kantarjian H, Pinto A, Schiffer CA, Nimer SD, Lowenberg B, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Wijermans PW, Gore S, Greenberg PL; World Health Organization(WHO) international working group. Report of an international working group to standardize response criteria for myelodysplastic syndromes. Blood. 2000 Dec 1;96(12):3671-4. PMID 11090046
- [Background] Cheson BD, Greenberg PL, Bennett JM, Lowenberg B, Wijermans PW, Nimer SD, Pinto A, Beran M, de Witte TM, Stone RM, Mittelman M, Sanz GF, Gore SD, Schiffer CA, Kantarjian H. Clinical application and proposal for modification of the International Working Group (IWG) response criteria in myelodysplasia. Blood. 2006 Jul 15;108(2):419-25. doi: 10.1182/blood-2005-10-4149. Epub 2006 Apr 11. PMID 16609072
- [Background] Parker JE, Mufti GJ. The myelodysplastic syndromes: a matter of life or death. Acta Haematol. 2004;111(1-2):78-99. doi: 10.1159/000074488. PMID 14646347
- [Background] Tehranchi R, Fadeel B, Forsblom AM, Christensson B, Samuelsson J, Zhivotovsky B, Hellstrom-Lindberg E. Granulocyte colony-stimulating factor inhibits spontaneous cytochrome c release and mitochondria-dependent apoptosis of myelodysplastic syndrome hematopoietic progenitors. Blood. 2003 Feb 1;101(3):1080-6. doi: 10.1182/blood-2002-06-1774. Epub 2002 Sep 5. PMID 12393561
- [Background] Tehranchi R, Invernizzi R, Grandien A, Zhivotovsky B, Fadeel B, Forsblom AM, Travaglino E, Samuelsson J, Hast R, Nilsson L, Cazzola M, Wibom R, Hellstrom-Lindberg E. Aberrant mitochondrial iron distribution and maturation arrest characterize early erythroid precursors in low-risk myelodysplastic syndromes. Blood. 2005 Jul 1;106(1):247-53. doi: 10.1182/blood-2004-12-4649. Epub 2005 Mar 8. PMID 15755901
- [Background] Tehranchi R, Fadeel B, Schmidt-Mende J, Forsblom AM, Emanuelsson E, Jadersten M, Christensson B, Hast R, Howe RB, Samuelsson J, Zhivotovsky B, Hellstrom-Lindberg E. Antiapoptotic role of growth factors in the myelodysplastic syndromes: concordance between in vitro and in vivo observations. Clin Cancer Res. 2005 Sep 1;11(17):6291-9. doi: 10.1158/1078-0432.CCR-04-1850. PMID 16144933
- [Background] Hellstrom-Lindberg E. Efficacy of erythropoietin in the myelodysplastic syndromes: a meta-analysis of 205 patients from 17 studies. Br J Haematol. 1995 Jan;89(1):67-71. doi: 10.1111/j.1365-2141.1995.tb08909.x. PMID 7833279
- [Background] Hellstrom-Lindberg E, Gulbrandsen N, Lindberg G, Ahlgren T, Dahl IM, Dybedal I, Grimfors G, Hesse-Sundin E, Hjorth M, Kanter-Lewensohn L, Linder O, Luthman M, Lofvenberg E, Oberg G, Porwit-MacDonald A, Radlund A, Samuelsson J, Tangen JM, Winquist I, Wisloff F; Scandinavian MDS Group. A validated decision model for treating the anaemia of myelodysplastic syndromes with erythropoietin + granulocyte colony-stimulating factor: significant effects on quality of life. Br J Haematol. 2003 Mar;120(6):1037-46. doi: 10.1046/j.1365-2141.2003.04153.x. PMID 12648074
- [Background] Remacha AF, Arrizabalaga B, Villegas A, Manteiga R, Calvo T, Julia A, Fernandez Fuertes I, Gonzalez FA, Font L, Junca J, del Arco A, Malcorra JJ, Equiza EP, de Mendiguren BP, Romero M. Erythropoietin plus granulocyte colony-stimulating factor in the treatment of myelodysplastic syndromes. Identification of a subgroup of responders. The Spanish Erythropathology Group. Haematologica. 1999 Dec;84(12):1058-64. PMID 10586205
- [Background] Jadersten M, Montgomery SM, Dybedal I, Porwit-MacDonald A, Hellstrom-Lindberg E. Long-term outcome of treatment of anemia in MDS with erythropoietin and G-CSF. Blood. 2005 Aug 1;106(3):803-11. doi: 10.1182/blood-2004-10-3872. Epub 2005 Apr 19. PMID 15840690
- [Background] Rigolin GM, Castoldi G. The role of rHuEpo in low-risk myelodysplastic syndrome patients. Leuk Lymphoma. 2005 Jun;46(6):823-31. doi: 10.1080/10428190500080348. PMID 16019526
- [Background] Casadevall N, Durieux P, Dubois S, Hemery F, Lepage E, Quarre MC, Damaj G, Giraudier S, Guerci A, Laurent G, Dombret H, Chomienne C, Ribrag V, Stamatoullas A, Marie JP, Vekhoff A, Maloisel F, Navarro R, Dreyfus F, Fenaux P. Health, economic, and quality-of-life effects of erythropoietin and granulocyte colony-stimulating factor for the treatment of myelodysplastic syndromes: a randomized, controlled trial. Blood. 2004 Jul 15;104(2):321-7. doi: 10.1182/blood-2003-07-2252. Epub 2004 Mar 30. PMID 15054036
- [Background] Herman JG, Baylin SB. Gene silencing in cancer in association with promoter hypermethylation. N Engl J Med. 2003 Nov 20;349(21):2042-54. doi: 10.1056/NEJMra023075. No abstract available. PMID 14627790
- [Background] Galm O, Herman JG, Baylin SB. The fundamental role of epigenetics in hematopoietic malignancies. Blood Rev. 2006 Jan;20(1):1-13. doi: 10.1016/j.blre.2005.01.006. Epub 2005 Feb 23. PMID 16426940
- [Background] Silverman LR, Demakos EP, Peterson BL, Kornblith AB, Holland JC, Odchimar-Reissig R, Stone RM, Nelson D, Powell BL, DeCastro CM, Ellerton J, Larson RA, Schiffer CA, Holland JF. Randomized controlled trial of azacitidine in patients with the myelodysplastic syndrome: a study of the cancer and leukemia group B. J Clin Oncol. 2002 May 15;20(10):2429-40. doi: 10.1200/JCO.2002.04.117. PMID 12011120
- [Background] Silverman LR, McKenzie DR, Peterson BL, Holland JF, Backstrom JT, Beach CL, Larson RA; Cancer and Leukemia Group B. Further analysis of trials with azacitidine in patients with myelodysplastic syndrome: studies 8421, 8921, and 9221 by the Cancer and Leukemia Group B. J Clin Oncol. 2006 Aug 20;24(24):3895-903. doi: 10.1200/JCO.2005.05.4346. PMID 16921040
- [Background] Kornblith AB, Herndon JE 2nd, Silverman LR, Demakos EP, Odchimar-Reissig R, Holland JF, Powell BL, DeCastro C, Ellerton J, Larson RA, Schiffer CA, Holland JC. Impact of azacytidine on the quality of life of patients with myelodysplastic syndrome treated in a randomized phase III trial: a Cancer and Leukemia Group B study. J Clin Oncol. 2002 May 15;20(10):2441-52. doi: 10.1200/JCO.2002.04.044. PMID 12011121
- [Background] Kaminskas E, Farrell A, Abraham S, Baird A, Hsieh LS, Lee SL, Leighton JK, Patel H, Rahman A, Sridhara R, Wang YC, Pazdur R; FDA. Approval summary: azacitidine for treatment of myelodysplastic syndrome subtypes. Clin Cancer Res. 2005 May 15;11(10):3604-8. doi: 10.1158/1078-0432.CCR-04-2135. PMID 15897554
- [Background] Cazzola M, Malcovati L. Myelodysplastic syndromes--coping with ineffective hematopoiesis. N Engl J Med. 2005 Feb 10;352(6):536-8. doi: 10.1056/NEJMp048266. No abstract available. PMID 15703418
- [Background] Musto P, Falcone A, Sanpaolo G, Bodenizza C, La Sala A, Perla G, Carella AM. Efficacy of a single, weekly dose of recombinant erythropoietin in myelodysplastic syndromes. Br J Haematol. 2003 Jul;122(2):269-71. doi: 10.1046/j.1365-2141.2003.04435.x. PMID 12846896
- [Background] Bowen D, Hyslop A, Keenan N, Groves M, Culligan D, Johnson P, Shaw A, Geddes F, Evans P, Porter J, Cavill I. Predicting erythroid response to recombinant erythropoietin plus granulocyte colony-stimulating factor therapy following a single subcutaneous bolus in patients with myelodysplasia. Haematologica. 2006 May;91(5):709-10. PMID 16670077
- [Background] 33. Mundle S, Lefebvre P, Duh MS, et al. Erythroid response (ER) rates in myelodysplastic syndromes (MDS) patients treated with epoetin alfa (EPO) or darbepoetin alfa (DARB) using International Working Group response criteria (IWGc): Comparative meta-analysis. Blood 2006; 108; 2672 (abstr
- [Background] Lyons RM, Cosgriff TM, Modi SS, Gersh RH, Hainsworth JD, Cohn AL, McIntyre HJ, Fernando IJ, Backstrom JT, Beach CL. Hematologic response to three alternative dosing schedules of azacitidine in patients with myelodysplastic syndromes. J Clin Oncol. 2009 Apr 10;27(11):1850-6. doi: 10.1200/JCO.2008.17.1058. Epub 2009 Mar 2. PMID 19255328
- See also: Spanish association of Haematology — http://www.aehh.org